CLINICAL TRIAL: NCT05954234
Title: Combining Pelvic Floor Rehabilitation With Postural Re-education in Women With Stress Urinary Incontinence and Chronic Low Back Pain: a Preliminary Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: I.R.C.C.S. Fondazione Santa Lucia (Other)
Responsible Party: Principal Investigator, Marco Tramontano, Head of Rehabilitation Services, I.R.C.C.S. Fondazione Santa Lucia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CE/PROG.593
Record Dates: First submitted 2023-04-07; First posted 2023-07-20 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Stress Urinary Incontinence; Low Back Pain
MeSH Terms: conditions — Urinary Incontinence, Stress; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pelvic floor rehabilitation and postural re-education (Active Comparator)
  Interventions: Other: Postural re-education; Other: Perineal Exercises
- pelvic floor rehabilitation and spinal mobilization (Active Comparator)
  Interventions: Other: Spinal mobilization; Other: Perineal Exercises

INTERVENTIONS:
Other: Postural re-education — Each session of the experimental approach will be composed of 40 minutes of postural exercise. Participants will be asked to maintain two different postures to stretch both the anterior and posterior muscle chains. The first posture will consist of lying on the back maintaining the extension of the legs to release the respiratory diaphragm and stretch the anterior muscle chain. For the second posture, participants wiil be asked to lie on their back with their legs flexed to stretch the posterior chai. For each posture, the physical therapist will use verbal commands and manual contact to maintain alignment and make the necessary postural corrections to optimize the stretching and discourage compensatory movements.
  10 sessions of the allocated intervention will be performed and organized in 2 times a week for 5 weeks.
  Arms: pelvic floor rehabilitation and postural re-education
Other: Spinal mobilization — This approach will consist of 40 minutes of thoracolumbar spine mobilization. Two different mobilizations will be carried out. In the first one the patient will be in sitting position with both legs out of the bed and a mobilization in antero-posterior direction will be provide by the physiotherapist; the second one will consist in rotational mobilisation provide with the patient in lateral decubitus position.
  10 sessions of the allocated intervention will be performed and organized in 2 times a week for 5 weeks.
  Arms: pelvic floor rehabilitation and spinal mobilization
Other: Perineal Exercises — Perineal Exercises will be performed in both the allocated approach. The protocol will consist in 10 minutes of perineal contraction and relaxation and 10 minutes of stretch-reflex for a total of 20 minutes of perineal exercises.10 sessions of the allocated intervention will be performed and organized in 2 times a week for 5 weeks.

SUMMARY:
Stress Urinary incontinence (SUI) is a common health condition in female population. Although its prevalence increases with the age, women of all ages could be affected. Several epidemiological studies have shown an association of SUI with Low Back Pain (LBP) demonstrating, moreover, that the presence of one condition may predispose the patient to the onset of the other. Concerning the LBP, the clinical practice guidelines provided recommendations for physical rehabilitative treatment. Different techniques and physical exercises have been developed and it is difficult at the date to affirm the superiority of one approach as compared to another. Moreover, the crucial role plays by the pelvic floor muscles (PFM) both as an integral part of trunk and lumbo-pelvic stability and in maintenance of urinary continence, lead the pelvic floor muscles disfunction to be associated both with SUI and LBP, making the PFM rehabilitation a useful approach in both the conditions. In this rehabilitative context the present study aims to verify the effectiveness of a global physical approach based on postural re-education combined to the pelvic floor rehabilitation in women with diagnosis of stress urinary incontinence associated with non-specific chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* woman aged from 18 to 75 years;
* diagnosis of Stress Urinary Incontinence associated with non-specific chronic Low Back Pain

Exclusion Criteria:

* severe pelvic organs prolapse (>second stage following the International Continence Society (ICS) classification);
* pregnancy;
* perineal denervation;
* inverted perineal command;
* presence of pelvic pain;
* fecal incontinence;
* vaginal infections;
* associated pathologies involving the Central Nervous System (CNS);
* psychotic disorders

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-20 (Actual); Primary Completion 2021-06-10 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
International Consultation on Incontinence Questionnaire-Urinary Short Form (ICIQ-UI SF) | Baseline, after after 5 weeks of treatment , and 1 month after the end of training
  Change of International Consultation on Incontinence Questionnaire-Urinary Short Form (ICIQ-UI SF) from baseline, at 10 sessions of treatment, and at 30 days after the end of the training. The ICIQ-UI SF evaluate the frequency, severity and impact on quality of life (QoL) of urinary incontinence. It is ranging from 0 to 21 where 0 is the minimum and 21 the maximum. An higer score indicates greater impairment from incontinence.

SECONDARY OUTCOMES:
Pain Visual Analogue Scale (VAS) | Baseline, after 5 weeks of treatment , and 1 month after the end of training
  Change of Pain Visual Analogue Scale (VAS) from baseline, at 10 sessions of treatment, and at 30 days after the end of the training. The VAS consisted in a straight horizontal line of fixed length (100 mm).
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100. A higher score indicates greater pain intensity.
Modified Oxford Scale (MOS) | Baseline, after 5 weeks of treatment , and 1 month after the end of training
  Change of Modified Oxford Scale (MOS) from baseline, at 10 sessions of treatment, and at 30 days after the end of the training. The MOS grading the patient's pelvic floot muscles' strength on a 0 to 5 scale, accordingly:
  0=No contraction
  1. =Flicker of movement
  2. =Through full range actively with gravity counterbalanced 3=Through full range actively against gravity 4=Through full range actively against some resistance 5=Through full range actively against strong resistance

CONTACTS AND LOCATIONS:
Locations (1):
- Marco Tramontano, Roma, Rm, Italy